CLINICAL TRIAL: NCT03486548
Title: Analgesic Efficacy of Adding SCB With Low Concentration Bupivacaine Combined With Dexamethasone to ACB and Periarticular Injection on Postoperative Pain After TKA: Randomized Controlled Study
Brief Title: Analgesic Efficacy of Adding SCB With Low Concentration Bupivacaine Combined With Dexamethasone on Pain After TKA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 768/2560(EC1)
Record Dates: First submitted 2018-03-15; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Total Knee Arthroplasty; Adductor Canal Block; Sciatic Nerve Block
Keywords: popliteal sciatic nerve block; total knee artgroplasty; adductor canal block; dexamethasone
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Lidocaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (Sham Comparator): adductor canal block with sham block
  Interventions: Drug: bupivacaine and lidocaine; Device: Ultrasound
- sciatic group (Experimental): adductor canal block with popliteal sciatic nerve block
  Interventions: Drug: bupivacaine and dexamethasone; Device: Ultrasound

INTERVENTIONS:
Drug: bupivacaine and dexamethasone — adductor canal block with 0.33% bupivacaine 15 ml with ultrasound guided popliteal sciatic block with 0.125% bupivacaine 20 ml and dexamethasone 5 mg
  Other Names: bupivacaine
  Arms: sciatic group
Drug: bupivacaine and lidocaine — adductor canal block with 0.33% bupivacaine 15 ml with ultrasound at popliteal sciatic area and subcutaneous infiltration popliteal area with 2% lidocaine 1 ml
  Arms: control group
Device: Ultrasound — ultrasound

SUMMARY:
This study evaluate the efficacy of adding popliteal sciatic nerve block with low concentration bupivacaine and dexamethasone to abductor canal block for total knee arthroplasty in patient with NSAIDs prescribing precaution. Half of participants will receive popliteal sciatic nerve block, abductor canal block and periarticular injection, while the other half will receive a sham block, abductor canal block and periarticular injection.

DETAILED DESCRIPTION:
After informed and consent, all patients will be devided into two groups, Sciatic group (group S) and Controlled group (group C). All patients will receive adductor canal block, then patients in group S will receive Sciatic nerve block with low concentration bupivacaine and dexamethasone while partients in group C will receive sham block. All patient will receive spinal anesthesia and intraoperative periarticular injection.

Postoperative pain score, muscle strength, total morphine consumption and adverse events will be record in case record form.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for single total knee arthroplasty
* patient with NSAIDs prescribing precautions such as history of NSAIDs allergy, Chronic kidney disease (GFR< 50 ml/min), history of ischemic heart disease or cerebrovascular disease

Exclusion Criteria:

* patient refusal
* body weight less than 45 kg
* history of allergy to bupivacaine or dexamethasone
* uncontrolled diabetes mellitus
* contraindicated for spinal block, adductor canal block or sciatic nerve block
* inability to assess pain score (cognitive or psychiatric history)
* patient scheduled for revision TKA
* preexisting neuropathy or neurological deficit in lower extremity
* preexisting chronic pain (prolonged use of oral morphine 20 mg/day or equivalent)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score at rest | postoperative 24 hours
  postoperative pain score at rest at 24 hour

SECONDARY OUTCOMES:
postoperative pain score at anterior and posterior site of knee | postoperative 24 hours
  postoperative pain score at anterior and posterior site of knee at 24 hour
postoperative pain score on 45 degree knee flexion and physical therapy | postoperative 24 hours
  postoperative pain score on 45 degree knee flexion and physical therapy
level of tibialis anterior muscle weakness | postoperative 24 hours
  level of tibialis anterior muscle weakness in 24 hour
adverse events | postoperative 24 hours
  perioperative adverse events such as LAST, hypotension, nausea and vomitting
total morphine consumption in postoperative 24 hours | postoperative 24 hours
  total morphine consumption in postoperative 24 hours
patient satisfaction | postoperative 24 hours
  patient satisfaction score
length of hospital stay | 7 days
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Busara Sirivanasandha, MD, Principal Investigator — Department of Anesthesia, Siriraj hospital, Mahidol university
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sirivanasandha B, Sutthivaiyakit K, Kerdchan T, Poolsuppasit S, Tangwiwat S, Halilamien P. Adding a low-concentration sciatic nerve block to total knee arthroplasty in patients susceptible to the adverse effects of non-steroidal anti-inflammatory drugs (NSAIDs): a randomized controlled trial. BMC Anesthesiol. 2021 Nov 13;21(1):282. doi: 10.1186/s12871-021-01491-7. PMID 34773995